

# Clinical Development

# Dabrafenib+Trametinib®

### DRB436B2205 / NCT02083354

Protocol 200104: An Open-Label, Multi-Center Study to Investigate the Objective Response Rate of Dabrafenib in Combination with Trametinib in Subjects with BRAF V600 Mutation-Positive Melanoma

# Statistical Analysis Plan (SAP)

Document type: SAP Documentation

Document status: Final

Release date: 05-May-2021

Number of pages: 39

00

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

# **Document History – Changes compared to previous final version of SAP**

| Date | Time point | Reason for update | Outcome<br>for<br>update | Section and title impacted (Current) |
|---|---|---|---|---|
| 11-<br>Aug-<br>2016 | Prior to DB lock | Creation of first version | First<br>version | NA |
| 06-<br>Apr-<br>2018 | Prior to DB lock | Creation of amendment 1 • Addition of PK samples for | Second<br>version | 2.9 |
| 2010 | | subjects with Day 1 or Day 15 samples | | 2.10 |
| | | <ul> <li>Revision of secondary<br/>objectives and endpoints in<br/>relation with the updated PK<br/>schedule</li> </ul> | | |
| | | • Update the RAP in line with Novartis RAP template | | |
| 05-<br>May- | Prior to<br>Final DB | Creation of final version for study closeout | Final version | 2.1 |
| 2021 | lock | • Specification of data included in the final analysis, remove the Pharmacokinetic analysis set | (for study closeout) | 2.2 |
| | | | | (PAS) which will not be used for the final analysis |
| | | • Remove details of Demographics, baseline characteristics, medical history, | | 2.4 |
| | | prior anti-cancer therapy,<br>Pharmacokinetic endpoint,<br>PD and PK/PD analyses, which | | 2.8 |
| | | will not change from the primary analysis | | 2.9 |
| | | • Remove the deails of overall compliance, Biomarkers analyses, since these analyses | | 2.10 |
| | | will not be included in the fianl CSR. | | 2.12 |
| | | • Simplify the sentences and remove some unplanned | | |

| Date | Time point | Reason for update | | | Outcome<br>for<br>update | Section and title impacted (Current) |
|---|---|---|---|---|---|---|
| | | analysis in section | Safety | analyses | | |

#### **Table of contents** Table of contents 4 List of abbreviations 6 1 1.1 1.2 Statistical methods 10 2.1 2.1.1 2.1.2 2.1.3 General definitions 11 2.2 2.2.1 Analysis Populations 13 2.2.2 2.2.3 2.3 Patient disposition \_\_\_\_\_\_\_14 2.3.1 2.3.2 Protocol deviations 14 2.3.3 Analysis sets 14 2.4 Treatments (study treatment, rescue medication, concomitant therapies, 2.4.1 2.4.2 2.5 2.5.1 2.5.2 2.5.3 Supportive analyses 20 2.5.4 2.6 2.7 Analysis of secondary efficacy objective(s)......20 2.7.1 2.7.2 Statistical hypothesis, model, and method of analysis......21 2.7.3 2.8 Safety analyses 23 2.8.1 Adverse events (AEs)......23 2.8.2 2.8.3

| | | 2.8.4 | Other safety data | 28 |
|---|---|---|---|---|
| | 2.9 | Pharma | acokinetic endpoints | |
| | 2.10 | PD and PK/PD analyses | | |
| | 2.11 | Patient- | -reported outcomes | 31 |
| | 2.12 | Biomar | kers | 31 |
| | | | | 31 |
| | 2.14 | Interim | analysis | 31 |
| 3 | Samp | le size ca | lculation | 31 |
| | 3.1 | Primary | y analysis | 31 |
| | 3.2 | Power | for analysis of key secondary variables | 31 |
| 4 | Chang | ge to prot | cocol specified analyses | 32 |
| 5 | | | | |
| | 5.1 | Imputat | tion rules | 33 |
| | | 5.1.1 | Study drug | 33 |
| | | 5.1.2 | AE, ConMeds and safety assessment date imputation | 34 |
| | | 5.1.3 | Other imputations | 35 |
| | 5.2 | AEs co | ding/grading | 36 |
| | 5.3 | Laborat | tory parameters derivations | 36 |
| | 5.4 | Statistic | cal models | 37 |
| | | 5.4.1 | Primary endpoint analysis | 37 |
| | | 5.4.2 | Secondary endpoint analysis | 38 |
| | 5.5 | Rule of | exclusion criteria of analysis sets | |
| 6 | Refer | | • | 38 |

#### List of abbreviations

AE Adverse event

ATC Anatomical Therapeutic Classification

AUC Area Under the Curve
bid bis in diem/twice a day
CR Complete Response
CSR Clinical Study report
CTC Common Toxicity Criteria

CTCAE Common Terminology Criteria for Adverse Events

DMC Data Monitoring Committee

DOR Duration of Response

eCRF Electronic Case Report Form

EOT End of Treatment FAS Full Analysis Set

HGRAC Human Genetic Resource Administration of China

IVR Interactive Voice Response
IWR Interactive Web Response

MedDRA Medical Dictionary for Drug Regulatory Activities

NCI National Cancer Institute

o.d. Once Daily

ORR Objective Response Rate

OS Overall Survival

PAS Pharmacokinetic Analysis Set

PD Progression Disease

PFS Progression-Free Survival

PK Pharmacokinetics
PPS Per-Protocol Set
PR Partial Response

PRO Patient-reported Outcomes qd Qua'que di'e / once a day

QoL Quality of Life

RECIST Response Evaluation Criteria in Solid Tumors

SAP Statistical Analysis Plan

SD Stable Disease
SOC System Organ Class
TFLs Tables, Figures, Listings
WHO World Health Organization

#### 1 Introduction

This statistical analysis plan (SAP) describes all planned analyses for the final Clinical Study Report (CSR) of study 200104 (DRB436B2205), a phase IIA, open label, multi-center study to investigate the objective response rate of Dabrafenib in combination with Trametinib in subjects with BRAF V600 mutation-positive melanoma.

The previous SAP for primary analysis was finalized on 06-Apr-2018, which described all planned analyses for the primary CSR. Based on the results in the primary CSR, dabrafenib and trametinib combination was approved in People's Republic of China (PRC).

This SAP is for the final analysis, i.e., the study closeout SAP. The content of this SAP is based on protocol DRB436B2205 Amendment v08. All decisions regarding final analysis, as defined in the SAP document, have been made prior to database lock of the study data.

# 1.1 Study design

This is a single-arm, Phase IIA, open-label, multi-center study evaluating safety and efficacy of dabrafenib and trametinib combination therapy in BRAF V600 mutant-positive melanoma.

Approximately 65 subjects were enrolled in the study.

Overall response rate (ORR), as assessed by local investigators review of tumor response and using RECIST 1.1 criteria, is the primary endpoint in this study.

The primary analysis was performed after all subjects had been followed for at least 16 weeks or had at least 2 tumor assessments or had discontinued study, with a data cut-off on 23-Feb-2018.

Treatment will continue until disease progression, death, unacceptable toxicity, or withdrawal of consent, or study completion. After treatment discontinuation, subjects will be followed for survival and disease progression as applicable.

Survival and new anti-cancer therapy follow-up will continue until study completion. The study completion is defined as:

- In case all subjects stop study treatment within 48 weeks after Last Subject First Visit (LSFV): the study is completed once the last subject has completed the 48 weeks survival follow-up or all subjects die or loss to follow-up, whichever comes first.
- In case some subjects are still on study treatment 48 weeks after LSFV: the study is completed once all subjects stop study medication, or all subjects who are still on study medication can have access to alternative supply of MEK/BRAF inhibitors, whichever comes first.

Doses of study treatment may be modified and/or interrupted for management of toxicities associated with study treatment.

No formal interim efficacy analysis is planned for this study.

# 1.2 Study objectives and endpoints

Table 1-1 Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To determine the objective response rate (ORR) of dabrafenib in combination with trametinib in subjects with BRAF V600 mutation-positive, unresectable or metastatic acral lentiginous or cutaneous melanoma | ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per RECIST v1.1 [Eisenhauer, 2009]. |
| Secondary | |
| To further evaluate the antitumor activity (progression-free survival (PFS), duration of response (DOR), and overall survival (OS)) | <ul> <li>PFS is defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.</li> <li>Duration of response is defined as the time from first documented evidence of CR or PR until the earliest date of documented radiological progression or death due to any cause among subjects who achieved a confirmed CR or PR.</li> <li>OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To assess exposures to dabrafenib, dabrafemetabolites, and trametinib after a single of and at steady-state, and characterize the population pharmacokinetics and pharmacodynamics of dabrafenib and trametinib | |
| To evaluate the safety and tolerability of<br>dabrafenib and trametinib | Safety as measured by clinical assessments including vital signs and physical examinations, 12-lead electrocardiograms (ECG), echocardiogram (ECHO), eye exams, chemistry and hematology laboratory values, and adverse events (AEs). |



#### 2 Statistical methods

# 2.1 Data analysis general information

SAS version 9.4 software will be used to perform all data analyses and to generate tables, figures and listings.

Data will be summarized following Novartis outputs shells, however data model will follow GSK legacy data (IDSL).

#### 2.1.1 Data included in the analysis

The Last Patient Last Visit (LPLV) date of the study is 19-Apr-2021, which will be used for final reporting (See section 1.1 for the definition of study completion).

Logically, all data collected in the database should be included in the final analysis and there should be no data cut-off. However, for Mainland Chinese patients, due to local regulations in China (lack of HGRAC approval), data from 01-Jul-2019 (inclusive) onwards can not be used, so there is a specific data cut-off of 30-Jun-2019 applied for these patients in this final analysis. For non Mainland Chinese patients, there is no data cut-off applied, i.e., all statistical analyses will be performed using all data collected in the database for these patients. All data with an assessment date or event start date (e.g. vital sign assessment date or start date of an adverse event) prior to or on the cut-off date will be included in the analysis. Any data collected beyond the cut-off date will not be included in the analysis and will not be used for any derivations.

All events with start date before or on the cut-off date and end date after the cut-off date will be reported as "ongoing". Events starting before or on the cut-off date and not having documented end date will be reported as "ongoing". This approach applies, in particular, to adverse event and concomitant medication reports. For these events, the end date will not be imputed and therefore will not appear in the listings.

# 2.1.2 General analysis conventions

**Pooling of centers:** Unless specified otherwise, data from all study centers will be pooled for the analysis. Due to expected small number of subjects enrolled at centers, no center effect will be assessed.

**Qualitative data** (e.g., gender, race, etc.) will be summarized by means of contingency tables by Mainland Chinese and all subjects; a missing category will be included as applicable. Percentages will be calculated using the number of subjects in the relevant population or subgroup as the denominator.

**Quantitative data** (e.g., age, body weight, etc.) will be summarized by appropriate descriptive statistics (i.e. mean, standard deviation, median, minimum, and maximum) by Mainland Chinese and all subjects.

Mainland Chinese population means the subjects enrolled from mainland China. All subjects means all subjects enrolled to the study.

#### 2.1.3 General definitions

### 2.1.3.1 Study drug and study treatment

Study drug and study treatment both refer to Dabrafenib in Combination with Trametinib.

# 2.1.3.2 Date of first/last administration of study drug

The date of first administration of study drug is defined as the first date when a non-zero dose of study drug is administered and recorded on the exposure form. For the sake of simplicity, the date of first administration of study drug will also be referred as start date of study drug.

The date of last administration of study drug is defined as the last date when a non-zero dose of study drug is administered and recorded on the exposure form. This date is also referred as last date of study drug.

#### 2.1.3.3 Study day

The study day for all assessments (e.g. tumor assessment, death, disease progression, tumor response, performance status, adverse event onset, laboratory abnormality occurrence, vital sign measurement, dose interruption) will be calculated using the start date of study drug as the origin. For assessments occurring after or on the start date of study drug, study day will be calculated as:

Study Day = Event date - start date of study drug + 1.

The first day of study drug is therefore study day 1.

For any assessment or events such as baseline disease characteristics or medical history (e.g., time since diagnosis of disease) occurring prior to the start of the study drug, study day will be negative and will be calculated as:

Study Day = Event date - start date of study drug.

The study day will be displayed in the data listings.

#### 2.1.3.4 Time unit

A year length is defined as 365.25 days. A month length is 30.4375 days (365.25/12). If duration is reported in months, duration in days will be divided by 30.4375. If duration is reported in years, duration in days will be divided by 365.25.

### **2.1.3.5** Baseline

Baseline will be defined as the most recent non-missing value prior to the first dose of study treatment. For laboratory data, baseline will be defined as the most recent non-missing value from a laboratory prior to the first dose of study treatment.

If subjects have no value as defined above, the baseline results will be considered missing.

# 2.1.3.6 On-treatment assessment/event and observation periods

For adverse event reporting the overall observation period will be divided into three mutually exclusive segments:

- 1. *pre-treatment period*: from day of subject's informed consent to the day before first administration of study treatment
- 2. *on-treatment period*: from date of first administration of study treatment to 30 days after date of last actual administration of any study treatment (including start and stop date)
- 3. *post-treatment period*: starting at day 31 after last administration of study treatment.

#### 2.1.3.7 Last contact date

The last contact date will be derived for subjects not known to have died at the analysis cut-off using the last complete date among the following:

Table 2-1 Last contact date data sources

| Source data | Conditions |
|---|---|
| Last contact date/last date subject was known to be alive from Survival Follow-up page | Subject status is reported to be alive |
| Start/End dates from further antineoplastic therapy | Non-missing medication/procedure term. |
| Start/End dates from drug administration record | Non-missing dose. Doses of 0 are allowed. |
| End of treatment date from end of treatment page | No condition. |
| Tumor (RECIST) assessment date | Evaluation is marked as 'done'. |
| Laboratory/PK collection dates | Sample collection marked as 'done'. |
| Vital signs date | At least one non-missing parameter value |
| Performance Status date | Non-missing performance status |

| Source data | Conditions |
|-----------------------|---------------------------|
| Start/End dates of AE | Non-missing verbatim term |

The last contact date is defined as the latest complete date from the above list on or before the data cut-off date. The cut-off date will not be used for last contact date, unless the subject was seen or contacted on that date. No date post cut-off date will be used. Completely imputed dates (e.g. the analysis cut-off date programmatically imputed to replace the missing end date of a dose administration record) will not be used to derive the last contact date. Partial date imputation is allowed for event (death)/censoring is coming from 'Survival information' eCRF.

The last contact date will be used for censoring of subjects in the analysis of overall survival.

# 2.2 Analysis sets

#### 2.2.1 Analysis Populations

#### **Full Analysis Set**

The Full Analysis Set (FAS) comprises all subjects to whom study treatment has been assigned and who received one dose of study treatment.

# **Safety Set**

The Safety Set includes all subjects who received any study treatment (i.e. at least one dose of any component of the study treatment).

FAS and Safety set are the same in this study.

#### 2.2.2 Withdrawal of Informed Consent

Any data collected in the clinical database after a subject withdraws informed consent from all further participation in the trial, will not be included in the analysis. The date on which a subject withdraws full consent is recorded in the eCRF.

Death events may be used in the analysis if captured from public records (registers), local law and subject informed consent permitting.

Additional data for which there is a separate informed consent, e.g. PK, biomarker etc., collected in the clinical database without having obtained that consent will not be included in the analysis.

### 2.2.3 Subgroup of interest

Not applicable

# 2.3 Patient disposition, demographics and other baseline characteristics

All demographic, other baseline disease characteristics and medical history data were summarized and listed during primary analysis, and therefore will not be summarized in the final analysis.

# 2.3.1 Patient disposition

Subject disposition information will be listed and summarized based on FAS. The number (%) of treated subjects included in the FAS will be presented. The number (%) of subjects in the FAS who discontinued the study and the reason for discontinuation will be presented by mainland Chinese and all subjects.

The following summaries will be provided (with % based on the total number of FAS subjects):

- Number (%) of subjects who are still on-treatment (based on the both dabrafenib and trametinib 'Study Treatment Discontinuation' pages not completed)
- Number (%) of subjects who discontinued the study treatment phase (based on both dabrafenib and trametinib 'Study Treatment Discontinuation' pages)
- Primary reason for study treatment phase discontinuation (based on dabrafenib or trametinib 'Study Treatment Discontinuation' pages)

In addition, the number (%) of subjects who have discontinued from the post-treatment follow-up and the reasons for discontinuation from the post-treatment follow-up will be provided.

#### 2.3.2 Protocol deviations

The number (%) of subjects in the FAS with protocol deviation will be tabulated by deviation category (as specified in the Protocol Deviation Management Plan) overall for the FAS. Major protocol deviations leading to exclusion from analysis sets will be tabulated separately by Mainland Chinese and all subjects. All the protocol deviations including the description will be listed.

The ongoing coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was first identified by the World Health Organization in Dec 2019. Since Mainland Chinese patients' data from 01-Jul-2019 onwards are not included in the final analysis due to local regulations in China, and there were no COVID-19 related PDs for other patients, thus COVID-19 related PDs are not considered.

#### 2.3.3 Analysis sets

The number (%) of subjects in each analysis set (defined in Section 2.2.1) will be summarized.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

### 2.4.1 Study treatment / compliance

### 2.4.1.1 Duration of study drug/treatment exposure

Extent of exposure to dabrafenib and trametinib will be summarized separately (see the details of duration of exposure below).

The duration of exposure to study treatment in months (from first day to last day of treatment) will be summarized. Descriptive statistics including mean, median, standard deviation, minimum, and maximum will be calculated for duration of exposure to study treatment. Moreover, duration of exposure to study treatment will be categorized in different time period: < 3 months, 3 months to 6 months, >6 months to 12 months, >12 months to 24 months, >24 months to 36 months and >36 months.

Duration of exposure to study treatment (days) = (last date of exposure to study treatment) – (date of first administration of study treatment) + 1.

The last date of exposure to study treatment is the last dates of exposure to investigational drug.

Duration of exposure by person time will be summarized by trametinib and dabrafenib. Person time of a specified group is defined as the total exposure time experienced by all subjects belonging to that specified group.

#### 2.4.1.2 Cumulative dose

Cumulative dose for any component of study treatment (dabrafenib or trametinib) is defined as the total dose given during the study treatment exposure.

The **planned cumulative dose** for a study treatment component refers to the total planned dose as per the protocol up to the last date of investigational drug administration.

The planned cumulative dose is not summarized/listed. It is used for relative dose intensity calculations.

The **actual cumulative dose** refers to the total actual dose administered, over the duration for which the subject is on the study treatment as documented in the Dose Administration eCRF.

For subjects who did not take any drug the cumulative dose is by definition equal to zero.

The subject daily dose, defined as the cumulative dose divided by the duration of exposure for each subject will be summarized.

Subject level listings of all doses administered on treatment along with dose change reasons will be produced.

The safety set will be used for all summaries and listings of study treatment.

#### 2.4.1.3 Dose intensity and relative dose intensity

The dose intensity (DI) and the relative dose intensity (RDI) for each study drug component (dabrafenib or trametinib) will be summarized by descriptive statistics. In addition, categorical

summary of RDI for each study drug component will be presented: <=75%, >75-90%, >90-110%, >110%.

**Dose intensity** (DI) for each study drug component in subjects with non-zero duration of exposure is defined as follows:

DI (dosing unit / day) = Actual Cumulative dose (dosing unit) / Duration of exposure to study treatment (day).

DI (mg/day) = Actual Cumulative dose (mg) / Duration of exposure (day)

For subjects who did not take any drug the DI is by definition equal to zero.

#### **Planned dose intensity** (PDI) is defined as follows:

PDI (dosing unit / day) = Planned Cumulative dose (dosing unit) / Duration of exposure (day).

Relative dose intensity (RDI) is defined as follows:

RDI = DI (dosing unit / day) / PDI (dosing unit / day).

DI and RDI will be summarized for each of the study treatment components.

The following tables provide the examples for the calculations, however, the final numbers should be based on the actual data, not from the following tables.

Table 2-2 Examples of dabrafenib dose administration and exposure

| DAR<br>record<br>number | Start/End<br>Date | Dose<br>Prescribed<br>(mg),<br>frequency | Dose<br>Administere<br>d (mg)<br>[total daily] | Dose<br>Changes,<br>Dose<br>Interruption | Dose<br>Permanently<br>Discontinued | Reason |
|---|---|---|---|---|---|---|
| 1 | 01Jan2016 /<br>05Jan2016 | 150 mg BID | 300 | No | No | |
| 2 | 06Jan2016 /<br>03Feb2016 | 150 mg BID | 200 | Yes | No | AE |
| 3 | 04Feb2016 /<br>25Feb2016 | 150 mg BID | 300 | No | No | |

Duration of exposure (days) = 25Feb2016 - 01Jan2016 + 1 = 56 days

Planned cumulative dose (for 56 days) = 300\*56 = 16800 mg

Actual cumulative dose = 300\*5 + 200\*29 + 300\*22 = 13900 mg

Dose intensity = 13900 mg / 56 days = 248.21 mg/day

Planned dose intensity = 16800 mg / 56 days = 300 mg/day

Relative dose intensity = DI / PDI = (248.21 mg/day) / (300 mg/day) = 0.83

Table 2-3 Examples of trametinib dose administration and exposure

| DAR<br>record<br>number | Start/End<br>Date | Dose<br>Prescribed<br>(mg),<br>frequency | Dose<br>Administere<br>d (mg)<br>[total daily] | Dose<br>Changes,<br>Dose<br>Interruption | Dose<br>Permanently<br>Discontinued | Reason |
|---|---|---|---|---|---|---|
| 1 | 01Jan2016 /<br>10Jan2016 | 2 QD | 2 | No | No | |
| 2 | 11Jan2016 /<br>15Jan2016 | 2 QD | 0 | Yes | No | AE |
| 3 | 16Jan2016 /<br>25Feb2016 | 1 QD | 1 | No | No | AE |

Duration of exposure = 25Feb2016 - 01Jan2016 + 1 = 56 days

Planned cumulative dose (for 56 days) = 2\*56 = 112 mg

Actual cumulative dose = 2\*10 + 0\*5 + 1\*41 = 61 mg

Dose intensity = 61 mg / 56 days = 1.09 mg/day

Planned dose intensity = 112 mg / 56 days = 2 mg/day

Relative dose intensity = DI / PDI = (1.09 mg/day) / (2 mg/day) = 0.54

#### 2.4.1.4 Dose reductions, interruptions or permanent discontinuations

The number of subjects who have dose reductions, permanent discontinuations or interruptions, and the reasons, will be summarized separately for each of the study treatment components.

'Dose interrupted', and 'Dose permanently discontinued' fields from the Study Treatment CRF pages (DAR) will be used to determine the dose reductions, dose interruptions, and permanent discontinuations, respectively.

The corresponding fields 'Reason for dose change/dose interrupted' and 'Reason for permanent discontinuation' will be used to summarize the reasons.

A dose change is either 'change in prescribed dose level' or 'dosing error' where actual dose administered/total daily dose is different from the prescribed dose.

For the purpose of summarizing interruptions and reasons, in case multiple entries for interruption that are entered on consecutive days with different reasons will be counted as separate interruptions. However, if the reason is the same in this mentioned multiple entries on consecutive days, then it will be counted as one interruption.

**Reduction**: A dose change where the prescribed dose level is lower than the previous prescribed dose level or where the actual dose administered/total daily dose is lower than the calculated dose amount based on the prescribed dose. Therefore any dose change to correct a dosing error will not be considered a dose reduction. Only dose change is collected in the CRF, number of reductions will be derived programmatically based on the change and the direction of the change.

A listing of actual treatments will be produced.

In addition, summaries of study treatment exposure and dose modifications (e.g. number of dose reductions, number of dose interruptions) will further characterize compliance. These analyses are described in Section 2.4.1

# 2.4.2 Prior, concomitant and post therapies

#### 2.4.2.1 Prior anti-cancer therapy

The number and percentage of subjects who received any prior anti-neoplastic medications, prior anti-neoplastic radiotherapy or prior anti-neoplastic surgery was summarized in primary analysis and therefore will not be summarized in the final analysis.

#### 2.4.2.2 Post treatment anti-cancer therapy

Anti-neoplastic therapies since discontinuation of study treatment will be listed and summarized by ATC class, preferred term, overall and by means of frequency counts and percentages using FAS.

#### 2.4.2.3 Concomitant medications

Concomitant therapy is defined as all interventions (therapeutic treatments and procedures) other than the study treatment administered to a subject coinciding with the study treatment period. Concomitant therapy include medications (other than study drugs) starting on or after the start date of study treatment or medications starting prior to the start date of study treatment and continuing after the start date of study treatment.

Concomitant medications will be coded using the World Health Organization (WHO) Drug Reference Listing (DRL) dictionary that employs the WHO Anatomical Therapeutic Chemical (ATC) classification system and summarized by lowest ATC class and preferred term using frequency counts and percentages. Surgical and medical procedures will be coded using MedDRA and summarized by SOC and preferred term. These summaries will include:

- 1. Medications starting on or after the start of study treatment but no later than 30 days after start of last dose of study treatment and
- 2. Medications starting prior to start of study treatment and continuing after the start of study treatment.

All concomitant therapies will be summarized. Any concomitant therapies starting and ending prior to the start of study treatment or starting more than 30 days after the last date of study treatment will be included. The safety set will be used for all concomitant medication tables and listings.

# 2.5 Analysis of the primary objective

The primary objective is to demonstrate the antitumor activity of dabrafenib in combination with trametinib as measured by ORR in subjects with BRAF V600 mutation-positive melanoma.

### 2.5.1 Primary endpoint

The primary endpoint, ORR is defined as the percentage of subjects, who have a confirmed complete response or a partial response based on RECIST 1.1 (Eisenhauer, 2009) and are evaluated by the investigator, among all subjects who have been enrolled and received at least one dose of investigational product. Tumor assessments performed before the start of any further antineoplastic therapy (i.e. any additional secondary antineoplastic therapy or surgery) will be considered in the assessment of overall response. Confirmation assessments must be performed no less than four weeks (28 days) after the criteria for response have initially been met and may be performed at the next protocol scheduled assessment. If a confirmation assessment is performed prior to the next protocol schedule assessment, the next protocol scheduled evaluation is still required.

ORR is defined as the proportion of subjects with confirm response of complete response (CR) or partial response (PR) according to RECIST 1.1. ORR will be calculated based on the FAS using local investigators review of tumor assessment data. Subjects with only non-measurable disease at baseline will be part of the analysis and will be included in the numerator only if a complete response was observed.

# 2.5.2 Statistical hypothesis, model, and method of analysis

The study will pursue an estimation strategy rather than formal hypothesis testing. This is reasonable given the proven performance of the combination therapy and the desire to estimate the effect in the Asian population. Since estimation is the goal, there are no formal hypotheses to be tested. 95% confidence limits for objective response rate (ORR) will be calculated. The minimal effect to be excluded from the lower end of the confidence interval for ORR will be 25%.

The primary objective was supported by the calculation of objective response rate using the FAS population. The primary analysis of ORR was performed after all enrolled subjects have completed 16 weeks of treatment or have at least 2 tumor assessments or have otherwise discontinued study treatment. The final analysis of ORR will be performed after LPLV.

The final efficacy analysis ORR will be summarized using descriptive statistics (N, %) along with 2-sided exact 95% confidence interval (CI) [Clopper and Pearson 1934].

#### 2.5.3 Handling of missing values/censoring/discontinuations

Subjects with unknown or missing response will be treated as non-responders, i.e. they will be included in the denominator when calculating the percentage. No imputation will be performed for missing lesion assessments or tumor response data.

Subjects with unknown or missing best overall response (BOR) will be counted as failures. If there is no baseline tumor assessment, all post-baseline overall lesion responses are expected to be 'Unknown'. If no valid post-baseline tumor assessments are available, the best overall response must be "Unknown" unless progression is reported. For the computation of ORR, these subjects will be included in the FAS and will be counted as 'failures'.

### 2.5.4 Supportive analyses

Not applicable

# 2.6 Analysis of the key secondary objective

There is no key secondary objective in this study.

# 2.7 Analysis of secondary efficacy objective(s)

The other secondary efficacy objectives are to describe PFS, OS, and DOR.

# 2.7.1 Secondary endpoints

Progression-Free Survival (PFS)

PFS is defined as the time from the date of the first dose to the date of the first documented progression or death due to any cause. PFS will be based on local investigators review of tumor assessments and using RECIST 1.1 criteria. The analysis will be based on FAS and will include all data observed up-to the cut-off date.

In the final analysis, PFS will be censored at the date of the last adequate tumor assessment if no PFS event is observed prior to the analysis cut-off date or before the start of the new anticancer therapy date or loss to follow up, whichever is earlier. (See Section 2.7.3 for additional details regarding censoring rules and determination of date of last adequate tumor assessment). Discontinuation due to disease progression (collected on the 'End of treatment' and 'End of post treatment follow up' disposition pages) without supporting objective evidence satisfying progression criteria per RECIST 1.1 will not be considered disease progression for PFS derivation. Clinical deterioration will not be considered as a qualifying event for progression for the final analysis.

Overall Survival (OS)

Overall Survival (OS) is defined as the time from date of first dose to date of death due to any cause. A cut-off date will be established for each analysis of OS. All deaths occurring on or before the cut-off date in the FAS will be used in the OS analysis.

If a subject is not known to have died at the time of analysis cut-off, OS will be censored at the date of last contact (See Section 2.1.1.7 for additional details). The survival distribution of OS distribution will be estimated using the Kaplan-Meier method, and Kaplan-Meier curves, medians and 95% confidence intervals of the medians intervals.

Duration of Response (DOR)

Duration of response (DOR) only applies to subjects whose confirmed overall response is complete response (CR) or partial response (PR) according to RECIST 1.1 based on local investigators review of tumor assessment data. The start date is the date of first documented response of CR or PR (i.e., the start date of response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death. Subjects continuing without progression or death due to underlying cancer will be censored at the date of their last adequate tumor assessment using the censoring rule described for PFS analysis (See Section 2.7.3 for additional details).

# 2.7.2 Statistical hypothesis, model, and method of analysis

Similar to the analysis of primary endpoint, there is no formal hypothesis testing. PFS, OS and DOR will be summarized descriptively using Kaplan-Meier medians and quartiles.

Since there is a single primary endpoint (ORR), supported by secondary endpoints, the nominal level of significance for the primary analysis will not be affected by multiplicity.

PFS based on local investigators review of tumor assessments and using RECIST 1.1 criteria is a secondary endpoint in this trial and will be analyzed using the same conventions as that of the primary efficacy analysis. The distribution of PFS will be estimated using the Kaplan-Meier method. The median PFS along with 95% confidence intervals will be presented.

The survival distribution of OS distribution will be estimated using the Kaplan-Meier method, and Kaplan-Meier curves, medians and 95% confidence intervals[Brookmeyer and Crowley 1982] of the medians intervals.

DOR will be listed and summarized for all subjects in the FAS with confirmed CR or PR. The distribution of duration of response will be estimated using the Kaplan-Meier method and the median duration of response will be presented along with 95% confidence interval only if a sufficient number of responses is observed.

# 2.7.3 Handling of missing values/censoring/discontinuations

For subjects who have not progressed or died at the time of the PFS or DOR analysis, censoring will be performed using the rules described in Table 2-4 or first dose for subjects without any adequate post baseline assessments.

PFS will be censored at the last adequate tumor assessment if one of the following occurs: absence of event; the event occurred after two or more missing tumor assessments. The term "missing adequate tumor assessment" is defined as a tumor assessment (TA) not performed or tumor assessment with overall lesion response of "UNK". The rule to determine number of missing TAs is based on the time interval between the date of last adequate tumor assessment and the date of an event. If the interval is greater than twice the protocol-specified interval between the TAs and 2 times the protocol-allowed time window around assessments, then the number of missing assessments will be 2 or more.

If there is no adequate baseline assessment, the subject will be censored at their date of the first dose. Subjects without any adequate post baseline tumor assessments will be censored at the date of the first dose. Subjects who progressed or died after an extended period without adequate assessment will be censored at their date of last adequate assessment prior to progression or death even if subsequent information is available regarding progression or death. An adequate assessment is defined as an assessment where the investigator determined response is CR, PR, or SD. The date of response at that assessment will be used for censoring. As the assessment schedule changes through the course of the protocol (i.e. every 8 weeks until week 56 and then every 12 weeks thereafter), the following rules will be used for identifying extended loss to follow up or extended time without an adequate assessment(i.e. two or more missed assessments).

• If death or PD is on or prior to day 399 (week 56 + 7 day window), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate

assessment during the time period of 119 days (16 weeks + 7 day window) prior to death or PD;

- Else if death or PD is after day 399 (week 56 + 7 day window) and prior to day 567 (week 80 + 7 day window), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate assessment during the time period of 147 days (8 weeks + 12 weeks + 7 day window) prior to death or PD.
- Else if death or PD is after day 567 (week 80 + 7 day window), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate assessment during the time period of 175 days (24 weeks + 7 day window) prior to death or PD.

For subjects who receive subsequent anti-cancer therapy the following rules will apply:

- If the start date of the anti-cancer therapy is partial (i.e. either missing the day but has the month and year available or missing both day and month), the imputation rules described in Section 5.1 will be applied. No imputation will be made for completely missing dates.
- If anti-cancer therapy is started without documented disease progression or is started prior to documented disease progression, then PFS will be censored at the date of the last adequate assessment that is no later than the date of initiation of anti-cancer
- therapy (i.e. if an assessment occurs on the same day as the start of new anti-cancer therapy the assessment will be used as it will be assumed the assessment occurred prior to the administration of new anti-cancer therapy). The date of response at the last adequate assessment will be used as the censoring date.
- If a subject has only a baseline visit or does not have an adequate assessment that is no later than the date of initiation of anti-cancer therapy, PFS will be censored at the date of the first dose

Refer to Table 2-4 for censoring and event date options and outcomes for PFS.

Table 2-3 Outcome and event/censor dates for PFS analysis

| Situation | Date | Outcome |
|---|---|---|
| No baseline assessment | Date of the first dose | Censored |
| Progression or death at or before next scheduled Assessment | Date of progression (or death) | Progressed |
| Progression or death after exactly one missing assessment | Date of progression (or death) | Progressed |
| Progression or death after two or more missing assessments | Date of last adequate assessment prior to missed assessment | Censored |
| No progression (or death) | Date of last adequate assessment | Censored |
| Treatment discontinuation due to 'Disease progression' without documented progression, i.e. | Date of last adequate assessment | Censored |

| Situation | Date | Outcome |
|---|---|---|
| clinical progression based on investigator claim | | |
| New anticancer therapy given prior to protocol defined progression | Date of last adequate<br>assessment on or prior to<br>starting new anti-cancer<br>therapy (or crossover<br>treatment) | Censored |
| Death before first PD assessment (including death at baseline or prior to any adequate assessments) | Date of death | Progressed |

# Overall survival (OS)

If a subject is not known to have died at the time of analysis cut-off, then OS will be censored at the date of last known date subject was alive, i.e., last contact date (see Table 2-1).

# 2.8 Safety analyses

All safety analyses will be based on the safety set.

# 2.8.1 Adverse events (AEs)

An overview summary of AEs, including counts and percentages of subjects with any AE, AEs related to study treatment, AEs leading to permanent discontinuation of study treatment, AEs leading to dose reductions, AEs leading to dose interruptions, AEs requiring additional therapy, SAEs, SAEs related to study treatment, fatal SAEs, and fatal SAEs related to study treatment will be produced.

A summary of non-serious AEs that occurred in strictly 5% of the subjects or above will be provided (no rounding for the percentage will be used in terms of 5% threshold, e.g. event with 4.9% incidence rate should not be included in this table). The summary will be displayed by SOC and PT. (for clinicaltrials.gov purpose)

AEs will be graded according to the CTCAE v4.0. Adverse events will be coded to the preferred term (PT) level using the Medical Dictionary for Regulatory Activities (MedDRA dictionary) (MedDRA 23.0).

A summary of number and percentage of subjects with any AE by maximum grade will be produced. AEs will be sorted by Preferred term (PT) in descending order of incidence. The summary will use the following algorithms for counting the subject:

- **Preferred term row**: Subjects experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- **Any event row**: Each subject with at least one adverse event will be counted only once at the maximum grade no matter how many events they have.

In addition, the number and percentage of AEs (all grades) will be summarized and displayed in two ways: 1) in descending order of incidence by PT only and 2) in descending order of

incidence by System Organ Classes (SOC) and PT. In the SOC row, the number of subjects with multiple events under the same system organ class will be counted once.

A separate summary will be provided for study treatment-related AEs. A study treatment-related AE is defined as an AE for which the investigator classifies the relationship to study treatment as "Yes". A worst case scenario approach will be taken to handle missing relatedness data, i.e. the summary table will include events with the relationship to study treatment as 'Yes' or missing. The summary table will be displayed in descending order of incidence by PT only.

All AEs will be listed. Additionally, a listing of subject IDs for each individual AE will be produced.

All SAEs will be tabulated based on the number and percentage of subjects who experienced the event. A summary will also be provided for study treatment-related SAEs. The summary tables will be displayed in descending order of incidence by PT only.

A study treatment-related SAE is defined as an SAE for which the investigator classifies the relationship to study treatment as "Yes". A worst case scenario approach will be taken to handle missing data, i.e. the summary table will include events with the relationship to study treatment as 'Yes' or missing.

SAEs are included in the listing of all adverse events. Separate supportive listings with subject-level details will be generated for all SAEs and Fatal SAEs.

AE summaries will include all AEs occurring during on-treatment period. All AEs collected in the AE (e)CRF page will be listed along with the information collected on those AEs e.g. AE relationship to study drug, AE outcome etc. AEs with start date outside of on-treatment period will be flagged in the listings.

AEs will be summarized by number and percentage of subjects having at least one AE, having at least one AE in each primary system organ class (SOC) and for each preferred term (PT) using MedDRA coding. A subject with multiple occurrences of an AE will be counted only once in the respective AE category. A subject with multiple CTCAE grades for the same preferred term will be summarized under the maximum CTCAE grade recorded for the event. AE with missing CTCAE grade will be included in the 'All grades' column of the summary tables

In AE summaries, the primary system organ class will be presented alphabetically and the preferred terms will be sorted within primary SOC in descending frequency. The sort order for the preferred term will be based on their frequency.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

If the same subject has more than one AE (irrespective of study treatment causality, seriousness and severity) with the same SOC and PT:

- a single occurrence will be counted if there is  $\leq 1$  day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted if there is > 1 day gap between the end date of the preceding AE and the start date of the consecutive AE

For legal requirements of clinicaltrials.gov (there is no requirement for EudraCT), the following two tables will be provided by system organ class and preferred term on the safety set population:

- On-treatment adverse events which are not SAEs with an incidence greater than and equal to 5%
- On-treatment deaths and SAEs suspected to be related to study treatment

# 2.8.1.1 Adverse events of special interest / grouping of AEs

An adverse event of special interest is a grouping of adverse events that are of scientific and medical concern specific to dabrafenib and trametinib. These groupings are defined using MedDRA terms, SMQs (standardized MedDRA queries), HGLTs (high level group terms), HLT (high level terms) and PTs (preferred terms). Customized SMQs (Novartis MedDRA queries, NMQ) may also be used. A NMQ is a customized group of search terms which defines a medical concept for which there is no official SMQ available or the available SMQ does not completely fit the need. It may include a combination of single terms and/or an existing SMQ, narrow or broad.

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of events.

All AE groupings for a clinical program are stored in the Compound Case Retrieval Strategy sheet (CRS) with clear versioning and reference to the MedDRA version used.

The events of special interest will be analysed using the most updated asset specific AESI (Adeverse Event of Special Interest) at the time of analysis.

For each specified AESI, number and percentage of subjects with at least one event of the AESI occurring during on treatment period will be summarized.

Summaries of these AESIs will be provided, (specifying grade, SAE, relationship, leading to treatment discontinuation, leading to dose adjustment/interruption, hospitalization, death, etc.). If sufficient number of events occurred, analysis of time to first occurrence will be applied.

A listing of all grouping levels down to the MedDRA preferred terms used to define each AESI will be generated.

#### 2.8.2 Deaths

In the event that a subject has withdrawn consent, no data after the withdrawal of consent date from this subject including death is supposed to appear in the database, which should be part of the data cleaning process.

All deaths occurring any time from the time of informed consent to the clinical cut-off date will be summarized based on the number and percentage of subjects. This summary will classify subjects by time of death relative to the last dose of medication (> 30 days or  $\leq$  30 days) and primary cause of death (disease under study, SAE related to study treatment, or other). A supportive listing will be generated to provide subject-specific details on subjects who died.

Separate summaries for on-treatment and all deaths (including post-treatment death) will be produced by system organ class and preferred term.

All deaths and deaths prior to starting treatment will be listed.

### 2.8.3 Laboratory data

The assessment of laboratory toxicities will examine the following laboratory tests:

**Hematology**: Hemoglobin (HGB), White Blood Cell (WBC) count, Total Neutrophils, Lymphocyte, Monocyte, Basophil and Eosinophil counts, and Platelet count. Basophils, Eosinophils and Monocytes are not gradable by CTCAE v4.0.

Clinical Chemistry: Sodium, Potassium, Calcium, Glucose, Blood Urea Nitrogen (BUN), Creatinine, Estimated Creatinine Clearance, Albumin, Lactate Dehydrogenase (LDH), and phosphate. BUN, LDH and Estimated Creatinine Clearance are not gradable by CTCAE v4.0. For Sodium, Potassium, Calcium, Phosphate, Lymphocyte and Glucose two bi-directional parameters (hyper and hypo), the tests will be graded by CTCAE v4.0 in both directions.

**Liver Function Tests**: Aspartate amino transferase (AST), Alanine amino transferase (ALT), Alkaline phosphatase, Total bilirubin (total) and Direct bilirubin. All these tests are gradable by CTCAE v4.0.

**Coagulation Tests**: Prothrombin time (PT) or International Normalized Ratio (INR), and partial thromboplastin time (PTT). These tests are collected only at baseline. Therefore these tests will not appear in any summaries of changes from baseline.

Summaries of worst case grade increase from baseline grade will be provided for all the lab tests that are gradable by CTCAE v4.0. These summaries will display the number and percentage of subjects with a maximum on-therapy grade increasing from their baseline grade. Any increase in grade from baseline will be summarized along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4. Missing baseline grade will be assumed as grade 0. In addition, the summary will include grade increase from baseline by scheduled visits. For laboratory tests that are graded for both low and high values, summaries will be done separately and labeled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by CTCAE v4.0, summaries of worst case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized at each scheduled visit as well as for the worst case post baseline. If a subject has a decrease to low and an increase to high during the same time interval, then the subject is counted in both the "Decrease to Low" categories and the "Increase to High" categories. Flag the earliest worst-case normal range values per time point. The worst-case for normal range values is bi-directional (either High or Low or both). If subject has both High and Low values in same time point, then flag both the earliest High record and the earliest Low record. If subject does not have a High or a Low value during the time point, then flag the subject's earliest in-range value. For visit timepoints: Baseline records are always flagged. Pre-therapy records, imputed records, and unscheduled records are not eligible for flagging.

Separate summary tables for (hematology, chemistry and liver function) laboratory tests will be produced.

Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value at each particular visit. For

subjects with a history of chronic Hepatitis B and/or Hepatitis C, the following tests will be performed at Screening:

- Viral hepatitis serology (HBs Antigen, HBc Antibody, HBs Antibody, HCV Antibody);
- Hepatitis BDNA; and/or
- Hepatitis C RNA.

As it is anticipated that the number of subjects with a history of chronic Hepatitis B and/or Hepatitis C will be small these data will only be listed and not summarized.

Summaries of hepatobiliary laboratory events including possible hy's law cases will be provided in addition to what has been described above.

On analyzing laboratory, data from all sources central and local laboratories will be combined. The summaries will include all assessments available for the lab parameter collected no later than 30 days after the last study treatment administration date.

The following summaries will be produced for hematology and biochemistry laboratory data (by laboratory parameter):

- Worst post-baseline CTC grade (regardless of the baseline status). Each subject will be counted only for the worst grade observed post-baseline.
- Shift tables using CTC grades to compare baseline to the worst on-treatment value
- For laboratory tests where CTC grades are not defined, shift tables using the low/normal/high/(low and high) classification to compare baseline to the worst ontreatment value.

The following listings will be produced for the laboratory data:

- Listings of all laboratory data, with CTC grades and classification relative to the laboratory normal range. Lab data collected during the post-treatment period will be flagged.
- Listing of all CTC grade 3 or 4 laboratory toxicities

#### **Liver function parameters**

Liver function parameters of interest are total bilirubin (TBL), ALT, AST and alkaline phosphatase (ALP). The number (%) of subjects with worst post-baseline values as per Novartis Liver Toxicity guidelines will be summarized:

The following summaries will be produced:

- ALT or AST > 3xULN
- ALT or AST > 5xULN
- ALT or AST > 8xULN
- ALT or AST > 10xULN
- ALT or AST > 20xULN
  - TBL > 2xULN
  - TBL > 3xULN
  - ALT or AST > 3xULN & TBL > 2xULN

ALT or AST > 3xULN & TBL > 2xULN & ALP < 2xULN (potential Hy's law)

Potential Hy's Law events are defined as those subjects with concurrent occurrence of AST or ALT > 3xULN and TBL > 2xULN and ALP < 2xULN in the same assessment sample during the on-treatment period. Further medical review has to be conducted to assess potential confounding factor such as, liver metastates, liver function at baseline etc.

# 2.8.4 Other safety data

### 2.8.4.1 ECG and cardiac imaging data

A summary of the number and percentage of subjects who had normal and abnormal (clinically significant and not clinically significant) ECG findings will be displayed by scheduled visits.

The QT and QTcB values based on Bazett formula will be rounded to the integer and the values will be categorized into the following ranges: Grade  $0 \leq 450$ , Grade  $1 \leq 450$  and 480, Grade  $2 \leq 480$  and 480, and Grade  $3 \leq 500$ . Summaries of grade increase will be provided. These summaries will display the number and percentage of subjects with any grade increase, increase to grade 480 and increase to grade 480 at each scheduled in the worst case post baseline only.

The changes in QT and QTcB values will be categorized into the clinical concern ranges which are specific to changes in QT and QTcB: (>30 and  $\le60$ ) and (>60) msec. A summary of change in QTcB value will display the number and percentage of subjects with a change within each range at each scheduled assessment time and in the worst case post baseline. Worst case post baseline will include both scheduled and unscheduled visits. Subjects with missing baseline values will be excluded from this summary.

The summaries for the QTcB will use the collected value based on Bazett formula. In addition, ECG interval values will be also be summarized.

Listings of abnormal ECG findings and a listing of ECG values will be provided.

LVEF Absolute change from baseline in LVEF will be summarized at each scheduled assessment time and in the worst case post baseline. Only the post baseline assessments that used the same method (ECHO or MUGA) as the baseline assessments will be used to derive the change from baseline. The change from baseline will be categorized as follows:

- Any increase
- No change
- Any decrease
  - >0 < 10 Decrease
    - 10 19 Decrease
  - >= 20 Decrease
- ≥10 decrease and ≥LLN
- >10 decrease and <LLN
- ≥20 decrease and ≥LLN
- >20 decrease and <LLN

LVEF results will also be listed with subject level details including absolute change from baseline.

Note: If there is any change in the methodology used throughout the study compared to baseline, the post-baseline values for which the methodology differs from baseline will be discarded in the tables presenting comparisons to baseline.

#### **Data handling**

In case the study requires ECG replicates at any assessment, the average of the ECG parameters at that assessment should be used in the analyses.

#### Data analysis

12-lead ECGs including QT, QTcB, and RR intervals will be obtained local for each subject during the study. ECG data will be read and interpreted locally

The number and percentage of subjects with notable ECG values will be presented.

- QT, QTcF, or QTcB
  - New value of > 450 and  $\le 480$  ms
  - New value of > 480 and  $\le 500$  ms
  - New value of > 500 ms
  - Increase from Baseline of  $> 30 \text{ ms to } \le 60 \text{ =ms}$
  - Increase from Baseline of > 60 ms
- RR
  - value < 600 ms
  - value  $\geq 600 \text{ ms}$

A listing of all ECG assessments will be produced and notable values will be flagged. A separate listing of only the subjects with notable ECG values may also be produced. In the listing, the assessments collected during the post-treatment period will be flagged.

#### 2.8.4.2 Vital signs

Vital sign assessments are performed in order to characterize basic body function. The following parameters were collected: height (cm), weight (kg), body temperature (°C), heart rate (beats per minute), systolic and diastolic blood pressure (mmHg).

#### Data handling

Vital signs collected on treatment will be summarized. Values measured outside of on treatment period will be flagged in the listings.

#### Data analysis

For analysis of vital signs the clinically notable vital sign criteria are provided in Table 2-5 below.

| Table 2-5 | Clinically | notable / | changes | in vital | signs |
|-----------|------------|-----------|---------|----------|-------|
| | • | | 0 | | 0.50 |

| Vital sign<br>(unit) | Clinically notable criteria | |
|---|---|---|
| | above normal value | below normal value |
| Weight (kg) | increase > 10% from Baseline | decrease > 10% from Baseline |
| Systolic blood pressure (mmHg) | >=180 with increase from baseline of >=20 | <=90 with decrease from baseline of >=20 |
| Diastolic blood<br>pressure<br>(mmHg) | >=105 with increase from baseline of >=15 | <=50 with decrease from baseline of >=15 |
| Pulse rate (bpm) | >=100 with increase from baseline of >25% | <=50 with decrease from baseline of > 25% |
| Body<br>temperature | >= 39.1 | |

The number and percentage of subjects with notable vital sign values (high/low) will be presented.

A listing of all vital sign assessments will be produced and notable values will be flagged. A separate listing of only the subjects with notable vital sign values may also be produced. In the listing, the assessments collected outside of on-treatment period will be flagged.

#### 2.8.4.3 Ophthalmic Examination

The ophthalmic examinations of tonometry will be listed.

### 2.8.4.4 Echocardiograms (ECHO)

Descriptive statistics of the left ventricular ejection fraction (LVEF) change and percent change from baseline to worst post-baseline value will be provided.

### 2.8.4.5 ECOG performance status

The ECOG PS scale (Table 2-6 will be used to assess physical health of subjects, ranging from 0 (most active) to 5 (least active):

Table 2-4 ECOG Performance Scale

| Score | Description |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |

| Score | Description |
|---|---|
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

Shift tables of ECOG performance status at baseline to worst post-baseline ECOG status by score will be provided. Shift tables of ECOG performance status at baseline to best post-baseline ECOG status by score will also be provided. ECOG performance status at each time point will be listed.

# 2.9 Pharmacokinetic endpoints

Not applicable for the final analysis as PK has already been analyzed and reported in the previous CSR, and no new PK data was collected since the primary analysis.

# 2.10 PD and PK/PD analyses

Not applicable.

# 2.11 Patient-reported outcomes

Not applicable.

#### 2.12 Biomarkers

Not applicable.



There is no interim analysis planned for this study.

# 3 Sample size calculation

# 3.1 Primary analysis

Approximately 65 subjects will be enrolled primarily based on clinical justification. This sample size was deemed to be sufficient to assess efficacy, safety and tolerability of Dabrafenib in combination with trametinib in Asian subjects with BRAF V600 Mutation-Positive Melanoma.

An exact binomial confidence interval will be calculated. Lower bound higher than 25% is considered to be clinically meaningful in this setting.

# 3.2 Power for analysis of key secondary variables

Not applicable.

# 4 Change to protocol specified analyses

Replace All Treated Subjects (ATS) to Full Analysis Set (FAS).

Mainland Chinese patients data from 01-Jul-2019 onwards are not included due to local regulations in China (lack of HGRAC approval).

# 5 Appendix

# 5.1 Imputation rules

In general imputed partial dates will not be used to derive study day, duration (e.g. duration of adverse events), or relapse time variables. In addition, imputed dates are not used for deriving the last contact date in overall survival analysis dataset.

#### 5.1.1 Study drug

The following rule should be used for the imputation of the dose end date for a given study treatment component:

**Scenario 1**: If the dose end date is completely missing and there is no EOT page and no death date, the subject is considered as on-going:

The subject should be treated as on-going and the cut-off date should be used as the dose end date.

**Scenario 2**: If the dose end date is completely or partially missing and the EOT page is available:

Case 1: The dose end date is completely missing, and the EOT completion date is complete, then this latter date should be used.

Case 2: Only Year(yyyy) of the dose end date is available and yyyy < the year of EOT date: Use Dec31yyyy

Case 3: Only Year(yyyy) of the dose end date is available and yyyy = the year of EOT date: **Use EOT date** 

Case 4: Both Year(yyyy) and Month (mm) are available for dose end date, and yyyy = the year of EOT date and mm < the month of EOT date:

### Use last day of the Month (mm)

Case 5: Both Year(yyyy) and Month (mm) are available for dose end date, and yyyy = the year of EOT date and mm = the month of EOT date:

#### **Use EOT date**

For subject with missing exposure end dates at the time of data cutoff, the exposure end date will be imputed to the earliest of: the date of the data cutoff, the date of withdrawal from the study, or the death date.

The imputed exposure end date will be used to calculate cumulative dose and exposure duration. The imputed exposure end date will be stored in the exposure analysis dataset and an exposure end date imputation flag variable will be derived indicating which exposure end date records are imputed. Imputed exposure end dates will also be stored on the study treatment end date variable.

For subjects who have missing end dates in their last exposure record because they are still on study treatment, the on-therapy indicator variables (time in relation to study treatment) are assigned to on-therapy for all records where the 'dataset'.'date' is after or on the study treatment start date. Missing exposure end date imputation will be applied to both study treatments (dabrafenib and trametinib). The study treatment end date variable will hold the last date of exposure across both study treatments.

All other cases should be considered as a data issue and the statistician should contact the data manager of the study.

After imputation, compare the imputed date with start date of treatment, if the imputed date is < start date of treatment:

#### Use the treatment start date

Subjects with missing start dates are to be considered missing for all study treatment component related calculations

# 5.1.2 AE, ConMeds and safety assessment date imputation

Table 5-1 Imputation of start dates (AE, CM) and assessments (LB, EG, VS)

| | T |
|---|---|
| Missing | Rule |
| Element | |
| day, month, and year | No imputation will be done for completely missing dates |
| day, month | <ul> <li>If available year = year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 01JanYYYY</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available year &gt; year of study treatment start date then 01JanYYYY</li> <li>If available year &lt; year of study treatment start date then 01JulYYYY</li> </ul> |
| Day | <ul> <li>If available month and year = month and year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 01MONYYYY.</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available month and year &gt; month and year of study treatment start date then 01MONYYYY</li> <li>If available month and year &lt; month year of study treatment start date then 15MONYYYY</li> </ul> |

Table 5-2 Imputation of end dates (AE, CM)

| Missing<br>Element | Rule (*=last treatment date plus 30 days provided it is not > (death date, cut-off date, withdrawl of consent date)) |
|---|---|
| day, month,<br>and year | <ul> <li>Completely missing end dates (incl. ongoing events) will be imputed by the end date of the on-treatment period*</li> <li>For post treatment period, no imputation will be done for completely missing dates</li> </ul> |
| day, month | • If partial end date contains year only, set end date = earliest of 31DecYYYY or end date of the on-treatment period * |

| Missing<br>Element | Rule (*=last treatment date plus 30 days provided it is not > (death date, cut-off date, withdrawl of consent date)) |
|---|---|
| | • For post treatment period, set end date = earliest of 31DecYYYY or death date or cut-off date or withdrawl of consent date |
| Day | <ul> <li>If partial end date contains month and year, set end date = earliest of last day of the month or end date of the on-treatment period*</li> <li>For post treatment period, set end date = earliest of last day of the month or death date or cut-off date or withdrawl of consent date</li> </ul> |
| Date of<br>progression<br>from Prior<br>anti-cancer<br>therapy | <ul> <li>Only impute when a month and year are available but the day is missing.</li> <li>Impute to last day of the month, also must be after the start date of therapy and prior to 'start of study treatment'. If 'start of study treatment ' is on the same month as prior therapy end date, then assign treatment start date minus one day for the prior therapy end date.</li> </ul> |

Any AEs and ConMeds with partial/missing dates will be displayed as such in the data listings.

Any AEs and ConMeds which are continuing as per data cut-off will be shown as 'ongoing' rather than the end date provided.

#### 5.1.3 Other imputations

#### Incomplete date of initial diagnosis of cancer and date of most recent recurrence

Missing day is defaulted to the 15<sup>th</sup> of the month and missing month and day is defaulted to 01-Jan.

#### Incomplete assessment dates for tumor assessment

All investigation dates (e.g. MRI scan, CT scan) must be completed with day, month and year. If one or more assessment dates are incomplete but other investigation dates are available, this/these incomplete date(s) are not considered for calculation of the assessment date and assessment date is calculated as the latest of all investigation dates (e.g. MRI scan, CT scan) if the overall response at that assessment is CR/PR/SD/UNK. Otherwise – if overall response is progression – the assessment date is calculated as the earliest date of all investigation dates at that evaluation number. If all measurement dates have no day recorded, the 1st of the month is used. If the month is not completed, for any of the investigations, the respective assessment will be considered to be at the date which is exactly between previous and following assessment. If a previous and following assessment is not available, this assessment will not be used for any calculation.

#### Applying the cut-off to tumor assessment

For tumor related assessments, if an evaluation has some assessments done prior to cut-off date and others after the cut-off date, then the evaluation is considered post-cut-off date and will be excluded from analysis.

# 5.2 AEs coding/grading

AEs will be graded according to the CTCAE v4.0. Adverse events will be coded to the preferred term (PT) level using the Medical Dictionary for Regulatory Activities (MedDRA dictionary)( MedDRA 23.0).

# 5.3 Laboratory parameters derivations

Grade categorization of lab values will be assigned programmatically as per NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The calculation of CTCAE grades will be based on the observed laboratory values only, clinical assessments will not be taken into account. The criteria to assign CTCAE grades are given in Novartis internal criteria for CTCAE grading of laboratory parameters. The latest available version of the document based on the underlying CTCAE version 4.0 at the time of analysis will be used. For laboratory tests where grades are not defined by CTCAE v4.0, results will be graded by the low/normal/high (or other project-specific ranges, if more suitable) classifications based on laboratory normal ranges.

A severity grade of 0 will be assigned for all non-missing lab values not graded as 1 or higher. Grade 5 will not be used. For laboratory tests that are graded for both low and high values, summaries will be done separately and labelled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia.

#### **Imputation Rules**

CTC grading for blood differentials is based on absolute values. However, this data may not be reported as absolute counts but rather as percentage of WBC.

If laboratory values are provided as '<X' (i.e. below limit of detection) or '>X', prior to conversion of laboratory values to SI unit, these numeric values are set to X.

The following rules will be applied to derive the WBC differential counts when only percentages are available for a xxx differential

```
xxx count = (WBC count) * (xxx %value / 100)
```

Further derivation of laboratory parameters might be required for CTCAE grading. For instance, corrected calcium can be derived using the reported total calcium value and albumin at the same assessment using the following formula:

Corrected Calcium (mg/dL) = Calcium (mg/dL) – 0.8 [Albumin (g/dL)-4]

In order to apply the above formula, albumin values in g/L will be converted to g/dL by multiplying by 0.1), calcium values in mmol/L will be converted to mg/dL by dividing by 0.2495. For calculation of laboratory CTC grades 0 and 1, the normal range for derived corrected calcium is set to the same limits (in mg/dL) as for calcium.

CTC grades for the derived absolute WBC differential counts (neutrophils, lymphocytes) and corrected calcium will be assigned as described above for grading

#### 5.4 Statistical models

# 5.4.1 Primary endpoint analysis

#### Overall response rate

Responses will be summarized in terms of percentage rates with 95% CIs. An exact binomial confidence interval (implemented using SAS procedure FREQ with EXACT statement) will be calculated [Clopper and Pearson 1934]

SAS procedure FREQ will be used to estimate the proportion of responders (binary outcome = 1 or "Yes"), along with the associated 95% (= $100 \times (1 - two\text{-sided alpha level})$ ) two-sided Pearson-Clopper CI.

Overall response will be determined using only target, non-target, and new lesions, using the criteria specified in the protocol.

Table 5-3 Evaluation of Overall Response for Subjects

| Target<br>Lesions | Non-Target Lesions | New Lesions | Overall Response |
|-------------------|---------------------|-------------|------------------|
| CR | CR or NA | No | CR |
| CR | Non-CR/Non-PD or NE | No | PR |
| PR | Non-PD or NA or NE | No | PR |
| SD | Non-PD or NA or NE | No | SD |
| NE | Non-PD or NA or NE | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

CR=complete response, PR = partial response, SD=stable disease, PD=progressive disease, NA= Not applicable, and NE=Not Evaluable

# **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression, death, or withdrawal of consent, whichever occurs first. Best overall response will be determined programmatically based on the investigator's assessment of response at each time point.

- To be assigned a status of SD, follow-up disease assessment must have met the SD criteria at least once after enrollment for a minimum of 49 days.
- If the minimum time for SD is not met, best response will depend on the subsequent assessments. For example, if an assessment of PD follows the assessment of SD and SD does not meet the minimum time requirement, the best response will be PD. Alternatively, subjects lost to follow-up after an SD assessment not meeting the minimum time criteria will be considered NE.

#### **Confirmation Criteria:**

- To be assigned a status of PR or CR, a confirmatory disease assessment should be performed no less than 4 weeks (28 days) after the criteria for response are first met.
- Confirmed best overall response will be determined programmatically based on RECIST 1.1.

# 5.4.2 Secondary endpoint analysis

# **Kaplan-Meier estimates**

An estimate of the survival function in each drug combination will be constructed using Kaplan-Meier (product-limit) method as implemented in PROC LIFETEST with METHOD=KM option. The PROC LIFETEST statement will use the option CONFTYPE=LOGLOG.

Median survival for each treatment drug combination will be obtained along with 95% confidence intervals calculated from PROC LIFETEST output using the method of [Brookmeyer and Crowley 1982]. Kaplan-Meier estimates of the survival function with 95% confidence intervals at specific time points will be summarized. The standard error of the Kaplan-Meier estimate will be calculated using Greenwood's formula.

Progression free survival will be using ONCTTE dataset and overall survival will be using ONCSURV dataset respectively.

# 5.5 Rule of exclusion criteria of analysis sets

Not applicable

#### 6 Reference

Eisenhauer EA, Therasse P, Bogaert J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-247.

Stein W, Yang J, Bates SE, Fojo T. Bevacizumab reduces growth rate constants of renal carcinomas: a novel algorithm suggests early discontinuation of bevacizumab resulted in a lack of survival advantage. Oncologist. 2008;13:1055-1062.

Wang Y, Sung, C, Dartois C, Ramchandani R, Booth BP, Rock E, et al. Elucidation of relationship between tumor size and survival in non-small cell lung cancer patients can aid early decision making in clinical drug development. Clin Pharmacol Ther. 2009;86:167-174.

Claret L, Girard P, Hoff PM, Van Cutsem E, Zuideveld KP, Jorga K, et al. Model-based prediction of phase III overall survival in colorectal cancer on the basis of phase II tumor dynamics. J Clin Oncol. 2009;27:4103-4108.

GlaxoSmithKline Document Number 2012N144949\_00 Study ID BRF113220. Population Pharmacokinetics and Exposure-Response Analysis of Dabrafenib and Trametinib in Combination. Report Date 17-Dec-2012.

Clopper CJ and Pearson PS, The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial, Biometrika, 1934, Vol. 26 (4) pp. 404-413

Brookmeyer R and Crowley J (1982). A Confidence Interval for the Median Survival Time. Biometrics, 38, 29 - 41.